CLINICAL TRIAL: NCT03896685
Title: Evaluating Newly Approved Drugs in Combination Regimens for Multidrug-Resistant TB With Fluoroquinolone Resistance (endTB-Q)
Acronym: endTB-Q
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Médecins Sans Frontières, France (Other)
Collaborators: Partners in Health (Other); Harvard Medical School (HMS and HSDM) (Other); Epicentre (Other); Institute of Tropical Medicine, Belgium (Other); Socios En Salud, Peru (Unknown); Interactive Research and Development (Other); University of San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSF ERB-1761
Record Dates: First submitted 2019-03-28; First posted 2019-04-01 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Tuberculosis, Multidrug-Resistant; Tuberculosis; Pulmonary Tuberculoses; Mycobacterial Infections; Bacterial Infections; Gram-Positive Bacterial Infections
Keywords: bedaquiline; delamanid; linezolid; clofazimine; tuberculosis; MDR-TB; XDR-TB
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant; Tuberculosis; Tuberculosis, Pulmonary; Mycobacterium Infections; Bacterial Infections; Gram-Positive Bacterial Infections; Extensively Drug-Resistant Tuberculosis | interventions — bedaquiline; OPC-67683; Tablets; Clofazimine; Linezolid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- endTB-Q: BeDeCLi 24 or 39 weeks (Experimental): endTB-Q regimen: bedaquiline-delamanid-linezolid-clofazimine (BeDeCLi). Subjects who are randomized to this arm will be assigned to duration of 24 or 39 weeks , according to the participant's extent-of-TB-disease phenotype. Participants may take as long as 32 weeks to complete all doses of a 24-week treatment regimen, and up to 47 weeks to complete all doses of a 39-week treatment regimen. Dosing of the experimental regimens will be oral and weight based.
  Interventions: Drug: Bedaquiline 100 MG; Drug: Delamanid 50 MG Oral Tablet; Drug: Clofazimine 100 MG Oral Capsule; Drug: Linezolid 600Mg Tab
- endTB-Q: Control arm (Active Comparator): endTB-Q is the control regimen, designed according to latest World Health Organization guidelines.
  Interventions: Drug: Control arm MDR-TB regimen, designed according to latest WHO guidelines

INTERVENTIONS:
Drug: Bedaquiline 100 MG — Bedaquiline: 400 mg QD x 2 weeks, followed by 200 mg 3x/week
  Other Names: TMC207
  Arms: endTB-Q: BeDeCLi 24 or 39 weeks
Drug: Delamanid 50 MG Oral Tablet — Delamanid: 100 mg BID
  Arms: endTB-Q: BeDeCLi 24 or 39 weeks
Drug: Clofazimine 100 MG Oral Capsule — Clofazimine: 100 mg QD
  Arms: endTB-Q: BeDeCLi 24 or 39 weeks
Drug: Linezolid 600Mg Tab — Linezolid: 600 mg QD up to Week 16, followed by 300 mg QD or 600 mg 3x/week according to a secondary randomization
  Arms: endTB-Q: BeDeCLi 24 or 39 weeks
Drug: Control arm MDR-TB regimen, designed according to latest WHO guidelines — Control arm MDR-TB regimen, designed according to latest WHO guidelines (might include bedaquiline, delamanid, linezolid, clofazimine, or all of these drugs).
  Arms: endTB-Q: Control arm

SUMMARY:
endTB-Q Clinical Trial is a Phase III, randomized, controlled, open-label, non-inferiority, multi-country trial evaluating the efficacy and safety of two new, all-oral, shortened regimens for multidrug-resistant tuberculosis (MDR-TB) with fluoroquinolone resistance.

DETAILED DESCRIPTION:
This is a Phase III, randomized, controlled, open-label, multi-country trial evaluating the efficacy of new combination regimens for treatment of fluoroquinolone-resistant MDR-TB.

Regimens examined combine newly approved drugs bedaquiline and delamanid with existing drugs known to be active against Mycobacterium tuberculosis (linezolid and clofazimine). The study will enroll in parallel across 1 experimental and 1 standard-of-care control arms, in a 2:1 ratio. Randomization will be stratified by country and extent-of-TB-disease phenotype. In the experimental arm, treatment will be for 24 or 39 weeks; duration will be assigned according to extent-of-TB-disease phenotype and treatment response. In the control arm, treatment will be delivered according to WHO guidelines (and local practice); duration will be variable. Trial participation in both arms will last at least until Week 73, and up to Week 104.

Non-inferiority will be established for the experimental arm if the lower bound of the one-sided 97.5% confidence interval around the difference in favorable outcome between the control and experimental arms is greater than or equal to -12%.

ELIGIBILITY:
Inclusion Criteria:

1. Has documented pulmonary tuberculosis due to strains of M. tuberculosis resistant to rifampin (RIF) and not susceptible to fluoroquinolones, according to a validated rapid molecular test. Patients with RIF-resistant TB who are unable to tolerate fluoroquinolones (history of severe adverse events, allergies, hypersensitivity) are also eligible, regardless of resistance/susceptibility to fluoroquinolones;
2. Is ≥15 years of age;
3. Is willing to use contraception: pre-menopausal women or women whose last menstrual period was within the preceding year, who have not been sterilized must agree to use contraception unless their partner has had a vasectomy; men who have not had a vasectomy must agree to use condoms;
4. Provides informed consent for study participation; additionally a legal representative of patients considered minor per local laws should also provide consent;
5. Lives in a dwelling that can be located by study staff and expects to remain in the area for the duration of the study.

Exclusion Criteria:

1. Has known allergies or hypersensitivity to any of the investigational drugs; 2. Is known to be pregnant or is unwilling or unable to stop breastfeeding an infant; 3. Is unable to comply with treatment or follow-up schedule; 4. Has any condition (social or medical) which, in the opinion of the site principal investigator, would make study participant unsafe; 5. a. Has had exposure (intake of the drug for 30 days or more) in the past five years to bedaquiline, delamanid, linezolid, or clofazimine, or has proven or likely resistance to bedaquiline, delamanid, linezolid, or clofazimine (e.g., household contact of a DR-TB index case who died or experienced treatment failure after treatment containing bedaquiline, delamanid, linezolid, or clofazimine or had resistance to one of the listed drugs); exposure to other anti-TB drugs is not a reason for exclusion.

b. Has received second-line drugs for 15 days or more prior to screening visit date in the current MDR/RR-TB treatment episode. Exceptions include:

1. patients whose treatment has failed according to the WHO definition and who are being considered for a new treatment regimen;
2. patients starting a new treatment regimen after having been "lost to follow-up" according to the WHO definition and,
3. patients in whom treatment failure is suspected (but not confirmed according to WHO definition), who are being considered for a new treatment regimen, and for whom the Clinical Advisory Committee (CAC) consultation establishes eligibility.

6. Has one or more of the following:

• Hemoglobin ≤7.9 g/dL;

• Uncorrectable electrolytes disorders:

* Total Calcium <7.0 mg/dL (1.75 mmol/L);
* Potassium <3.0 mEq/L (3.0 mmol/L) or ≥6.0 mEq/L (6.0 mmol/L);
* Magnesium <0.9 mEq/L (0.45 mmol/L);

  * Serum creatinine >3 x ULN;
  * Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) ≥3 x ULN;
  * Total bilirubin ≥3 x ULN; Unless otherwise specified, Grade 4 result as defined by the MSF Severity Scale on any of the screening laboratory tests.

    7. Has cardiac risk factors defined as:
  * An arithmetic average of the two ECGs with highest QTcF intervals of greater than or equal to 450 ms. Retesting to reassess eligibility will be allowed using an unscheduled visit during the screening phase;
  * Evidence of ventricular pre-excitation (e.g., Wolff Parkinson White syndrome);
  * Electrocardiographic evidence of either:
* Complete left bundle branch block or right bundle branch block; OR
* Incomplete left bundle branch block or right bundle branch block and QRS complex duration greater than or equal to 120 msec on at least one ECG; • Having a pacemaker implant;

  * Congestive heart failure;
  * Evidence of second or third degree heart block;
  * Bradycardia as defined by sinus rate less than 50 bpm;
  * Personal or family history of Long QT Syndrome;
  * Personal history of arrhythmic cardiac disease, with the exception of sinus arrhythmia;
  * Personal history of syncope (i.e. cardiac syncope not including syncope due to vasovagal or epileptic causes).

    8. Concurrent participation in another trial of any medication used or being studied for TB treatment, as defined in cited documents.

    9. Is taking any medication that is contraindicated with the medicines in the trial regimen which cannot be stopped (with or without replacement) or requires a wash-out period longer than 2 weeks.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2020-04-06 (Actual); Primary Completion 2024-10-04 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Week 73 Efficacy: Proportion of participants with favorable outcome at Week 73 | Week 73 after randomization
  Proportion of participants with favorable outcome at Week 73. A participant's outcome will be classified as favorable at Week 73 if the outcome is not classified as unfavorable, and one of the following is true:
  1. The last two culture results are negative. These two cultures must be taken from sputum samples collected on separate visits, the latest between Week 65 and Week 73;
  2. The last culture result (from a sputum sample collected between Week 65 and Week 73) is negative; and either there is no other post-baseline culture result or the penultimate culture result is positive due to laboratory cross contamination; and bacteriological, radiological and clinical evolution is favorable;
  3. There is no culture result from a sputum sample collected between Week 65 and Week 73 or the result of that culture is positive due to laboratory cross contamination; and the most recent culture result is negative; and bacteriological, radiological and clinical evolution is favorable.

SECONDARY OUTCOMES:
Week 104 Efficacy: Proportion of participants with favorable outcome at Week 104 | Week 104 after randomization
  Proportion of participants with favorable outcome at Week 104. A participant's outcome will be classified as favorable at Week 104 if the outcome is not classified as unfavorable, and one of the following is true:
  1. The last two cultures are negative. These two cultures must be from sputum samples collected on separate visits, the latest between Week 97 and Week 104;
  2. The last culture result (from a sputum sample collected between Week 97 and Week 104) is negative; and either there is no other post-baseline culture result or the penultimate culture result is positive due to laboratory cross contamination; and bacteriological, radiological and clinical evolution is favorable;
  3. There is no culture result from a sputum sample collected between Week 97 and Week 104 or the result of that culture is positive due to laboratory cross contamination; and the most recent culture result is negative; and bacteriological, radiological and clinical evolution is favorable.
Early Treatment Response (culture conversion) | Week 8 after randomization
  1. Proportion of patients with culture conversion assessed in MGIT system (and LJ where possible): 2 consecutive negative cultures from specimens collected at 2 different visits; if there is a missing or contaminated culture between 2 negatives, the definition of conversion is still met;
  2. Time to culture conversion: assessed in MGIT system (and LJ where possible): time from treatment initiation to first of 2 consecutive negative cultures; if there is a missing or contaminated culture between 2 negatives, the definition of conversion is still met;
  3. Change in time to positivity (TTP) in MGIT over first 8 weeks.
Week 39 Efficacy: Proportion of participants with favorable outcome at Week 39 | Week 39 after randomization
  Proportion of participants with favorable outcome at Week 39. A participant's outcome will be classified as favorable at Week 39 if all culture results from samples collected between Week 36 and Week 39 are negative and the outcome is not classified as unfavorable.
  A participant's outcome will be classified as unfavorable at Week 39 in case of:
  1. In the experimental arm, addition or replacement of one or more drugs;
  2. In the control arm, addition or replacement of two or more drugs;
  3. Death from any cause;
  4. At least one culture result (from a sample collected between Week 36 and Week 39) is positive;
  5. The patient is not assessable because the last available culture result is from a sample collected before Week 36;
Week 73 Failure/Relapse | Week 73 after randomization
  Proportion of participants with treatment failure/relapse. A participant's outcome will be classified as failure/relapse at Week 73 if:
  1. In an experimental arm, addition or replacement of one or more drugs;
  2. In the control arm, addition or replacement of two or more drugs;
  3. Initiation of a new MDR-TB regimen after the end of the allocated study regimen and before Week 73;
  4. At least one of the last two cultures, the latest between Week 65 and 73, is positive in the absence of cross contamination;
  5. The last culture result between Week 65 and 73 is negative; and: there is no other post-baseline culture result or the penultimate culture is positive due to cross contamination; and bacteriological, radiological or clinical evolution is unfavorable;
  6. There is no culture result between Week 65 and 73 or it is positive due to cross contamination; and: the most recent culture is negative; and bacteriological, radiological or clinical evolution is unfavorable.
Week 104 Failure/Relapse | Week 104 after randomization
  Proportion of participants with treatment failure/relapse. A participant's outcome will be classified as failure/relapse at Week 104 if:
  1. In an experimental arm, addition or replacement of one or more drugs;
  2. In the control arm, addition or replacement of two or more drugs;
  3. Initiation of a new MDR-TB treatment regimen after the end of the allocated study regimen and before Week 104;
  4. At least one of the last two cultures, the latest between Week 97 and 104, is positive in the absence of cross contamination;
  5. The last culture result between Week 97 and 104 is negative; and: there is no other post-baseline culture result or the penultimate culture is positive due to cross contamination; and bacteriological, radiological or clinical evolution is unfavorable;
  6. There is no culture result between Week 97 and 104 or it is positive due to cross contamination; and: the most recent culture is negative; and bacteriological, radiological or clinical evolution is unfavorable.
Week 73 Survival | Week 73 after randomization
  At 73 weeks, the proportion of patients who died of any cause
Week 104 Survival | Week 104 after randomization
  At 104 weeks, the proportion of patients who died of any cause
Week 73 AEs and SAEs | Week 73 after randomization
  The proportion of participants with grade 3 or greater AEs and serious adverse events (SAEs) of any grade by 73 weeks
Week 104 AEs and SAEs | Week 104 after randomization
  The proportion of participants with grade 3 or greater AEs and serious adverse events (SAEs) of any grade by 104 weeks
Week 73 AESIs | Week 73 after randomization
  The proportion of participants with adverse events of special interest (AESIs) by 73 weeks
Week 104 AESIs | Week 104 after randomization
  The proportion of participants with adverse events of special interest (AESIs) by 104 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Guglielmetti, MD, Principal Investigator — Médecins Sans Frontières, France; Carole Mitnick, Sc.D, Principal Investigator — Harvard Medical School (HMS and HSDM)
Locations (10):
- Aundh Chest Hospital, Pune, India
- Kazakhstan (2):
  - National Center for Tuberculosis Problems, Almaty
  - State Municipal Enterprise on the right of economic management "City Centre of Phthisiopulmonology" of Nur-sultan city's administration, Almaty
- Partners In Health Lesostho, Maseru, Lesotho
- Pakistan (2):
  - The Indus Hospital, Karachi
  - Institute of Chest Disease,, Kotri
- Peru (2):
  - Centro de Investigación del Hospital Nacional Hipólito Unanue, Lima
  - Centro de Investigación de Enfermedades Neumológicas del Hospital Nacional Sergio Bernales, Lima
- Vietnam (2):
  - Hanoi Lung Hospital, Hanoi
  - Pham Ngoc Thach Hospital, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
After deidentification process most part of variables recorded in the eCRF (no patients name or ID, no site or country location, no dates but intervals from randomization, no birth dates but age at randomization, no information on staff...).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: From 2025 end and will last 4 years renewable.
Access Criteria: * proposal has scientific value / the scientific question addresses a knowledge gap and avoids duplication without added value and unnecessary competition, and benefits the wider public health community
  * the data requested must be capable of answering the research question, and each variable requested must be required for the successful completion of the research
  * the methodology proposed to answer the research question must be sound
  * conform to the Data Access Guidelines, Ethics Framework, and Conflict of Interest Policy (see on website https://endtb.org/data-sharing-initiative)
URL: http://endtb.org/data-sharing-initiative

REFERENCES:
- [Derived] Guglielmetti L, Khan U, Velasquez GE, Gouillou M, Ali MH, Amjad S, Kamal F, Abubakirov A, Ardizzoni E, Baudin E, Bektassov S, Berry C, Bonnet M, Chavan V, Coutisson S, Dakenova Z, de Jong BC, Dinh LV, Ferlazzo G, Kirakosyan O, Lachenal N, Lecca L, McIlleron H, Mikanda KK, Mucching-Toscano S, Mulders W, Mushtaque H, Nahid P, Nguyen DV, Nguyen NV, Oyewusi L, Motta I, Panda S, Patil S, Pham TH, Phan DT, Phan HTT, Phillips PPJ, Ruiz J, Rupasinghe P, Salahuddin N, Sanchez-Garavito E, Seung KJ, Asfaw MT, Vargas Vasquez D, Rich ML, Varaine F, Mitnick CD; endTB-Q Clinical Trial Team. Bedaquiline, delamanid, linezolid, and clofazimine for rifampicin-resistant and fluoroquinolone-resistant tuberculosis (endTB-Q): an open-label, multicentre, stratified, non-inferiority, randomised, controlled, phase 3 trial. Lancet Respir Med. 2025 Sep;13(9):809-820. doi: 10.1016/S2213-2600(25)00194-8. Epub 2025 Jul 16. PMID 40683298
- [Derived] Patil SB, Tamirat M, Khazhidinov K, Ardizzoni E, Atger M, Austin A, Baudin E, Bekhit M, Bektasov S, Berikova E, Bonnet M, Caboclo R, Chaudhry M, Chavan V, Cloez S, Coit J, Coutisson S, Dakenova Z, De Jong BC, Delifer C, Demaisons S, Do JM, Dos Santos Tozzi D, Ducher V, Ferlazzo G, Gouillou M, Khan U, Kunda M, Lachenal N, LaHood AN, Lecca L, Mazmanian M, McIlleron H, Moreau M, Moschioni M, Nahid P, Osso E, Oyewusi L, Panda S, Paquet A, Thuong Huu P, Pichon L, Rich ML, Rupasinghe P, Salahuddin N, Sanchez Garavito E, Seung KJ, Velasquez GE, Vallet M, Varaine F, Yuya-Septoh FJ, Mitnick CD, Guglielmetti L. Evaluating newly approved drugs in combination regimens for multidrug-resistant tuberculosis with fluoroquinolone resistance (endTB-Q): study protocol for a multi-country randomized controlled trial. Trials. 2023 Nov 30;24(1):773. doi: 10.1186/s13063-023-07701-6. PMID 38037119

DOCUMENTS (6):
  • Informed Consent Form: endTB-Q_Research Screening Adult Consent_Assent form V4.3 (2022-07-05): https://cdn.clinicaltrials.gov/large-docs/85/NCT03896685/ICF_006.pdf
  • Informed Consent Form: endTB-Q_Research Screening Parental Consent form V4.3 (2022-07-05): https://cdn.clinicaltrials.gov/large-docs/85/NCT03896685/ICF_007.pdf
  • Informed Consent Form: endTB-Q_Research Adult Consent_Assent form v4.3 (2022-07-05): https://cdn.clinicaltrials.gov/large-docs/85/NCT03896685/ICF_008.pdf
  • Informed Consent Form: endTB-Q_Research Parental Consent form v4.3 (2022-07-05): https://cdn.clinicaltrials.gov/large-docs/85/NCT03896685/ICF_009.pdf
  • Informed Consent Form: endTB-Q_Pregnant Partner Consent form V4.3 (2022-07-05): https://cdn.clinicaltrials.gov/large-docs/85/NCT03896685/ICF_010.pdf
  • Informed Consent Form: endTB-Q_Treatment during pregnancy_Consent form V4.3 (2022-07-05): https://cdn.clinicaltrials.gov/large-docs/85/NCT03896685/ICF_011.pdf